CLINICAL TRIAL: NCT03250845
Title: Comparison of Multigam IV (5% vs. 10%) as Substitution Therapy in Patients With an Immunodeficiency Secondary to a Hematological Disorder to Evaluate Infusion Time, Tolerance and Satisfaction. A Monocentric Observational Belgian Study
Brief Title: Comparison of Multigam IV (5% vs. 10%) in Patients With an Immunodeficiency Secondary to a Hematological Disorder
Acronym: MULTISIM
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: HEM-2017-001
Record Dates: First submitted 2017-08-07; First posted 2017-08-16 (Actual); Results first posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-10

CONDITIONS: Hematologic Diseases; Secondary Immune Deficiency
Keywords: Multigam; Immunoglobulin; Secondary immunodeficiency
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this observational study is to compare the administration of standard of care Multigam IV 5% and standard of care Multigam IV 10% in order to observe changes in infusion time and infusion related reactions. Patient satisfaction, number of actions taken by the nursing staff during infusion and satisfaction of the nursing staff will also be evaluated.

DETAILED DESCRIPTION:
Given the growing number of patient contacts at our day-care center, there is a continuous search to further improve the flow and to shorten the time spent per patient at the day-care center, without loss of quality in care.

In order to achieve this goal, this study wants to compare the administration of Multigam IV 5% and Multigam IV 10%. Multigam 5% and Multigam 10% are immunoglobulin solutions that are administered to strengthen the body's natural defense system (immune system). In case of recurrent infections, patients with an immunodeficiency secondary to a hematologic disorder can be treated with immunoglobulin substitution therapy. Patients can receive Multigam IV 5% and Multigam IV 10% in daily clinical practice and will receive both formulations in the same manner and intensity, meaning their use is not limited to this study.

For this observational study, patients with an immunodeficiency secondary to a hematologic disorder will be evaluated for inclusion. Patient characteristics, infusion time, time spent at the day-care center, adverse events and number of actions taken by the nursing staff will be evaluated for Multigam 5% administration. After 3-4 weeks, patients will return for Multigam 10% administration and an identical evaluation will take place along with a questionnaire for the patient and nursing staff to assess their satisfaction. The results will be processed to compare and evaluate the administration of both immunoglobulin solutions.

ELIGIBILITY:
Inclusion Criteria:

* Age => 18 years
* Immunodeficiency secondary to a hematologic disorder
* Patient has received at least 2 Multigam IV 5% administrations
* Patient may not have had any adverse events (grade 2 or higher according to CTCAE v4.03) during the last 2 Multigam IV 5% administrations
* Patient needs at least 2 more immunoglobulin administrations
* Signed informed consent

Exclusion Criteria:

* Patient has received less than 2 Multigam IV 5% administrations
* Patient has had an adverse event (grade 2 or higher according to CTCAE v4.03) during the last 2 Multigam IV 5% administrations
* Refusal to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients with an immunodeficiency secondary to a hematologic disorder
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Delforge, MD PhD, Principal Investigator — UZ Leuven Gasthuisberg
Locations (1):
- UZ Leuven Gasthuisberg, Leuven, Vlaams-Brabant, Belgium

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled 30 patients with an immunodeficiency secondary to a hematologic disorder requiring immunoglobin substitution therapy from 1 academic center in Belgium. The last patient completed in December 2017.
Groups:
- All Study Participants: 30 participants who received Multigam 5% intravenous immunoglobulin (IVIg) and Multigam 10% intravenous immunoglobulin (IVIg) 3 to 4 weeks later.
  Dosing was set at 0.4 g/kg for both infusions.
Period: Multigam 5% Infusion (Baseline)
Arm/Group | All Study Participants
Started | 30
Completed | 30
Not Completed | 0
Period: Multigam 10% Infusion (3-4 Weeks Later)
Arm/Group | All Study Participants
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Baseline characteristics of the study population (30 participants).
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 30
Haematological disorder [Count of Participants; unit: Participants]
  Plasma Cell Dyscrasia: Scleromyxedema | 1
  AL Amyloidosis | 2
  Multiple Myeloma | 12
  Chronic Lymphocytic Leukemia | 9
  Diffuse Large B-Cell Lymphoma | 2
  Follicular Lymphoma | 2
  Non-Hodgkin Lymphoma, Unclassifiable | 2
Time between first IVIg infusion and start of study [Mean (Standard Deviation); unit: years] | 4.1 (4.3)
First Multigam Dosage [Median (Full Range); unit: gram] | 30 [20 to 70]

OUTCOME MEASURES:

1. Primary Outcome: Infusion Time of Multigam IV 5% and Multigam IV 10%
Description: Comparison of infusion time between Multigam (MG) IV 5% and Multigam IV 10%. Results will be assessed by Student's-t-test and 95% confidence interval.
Time Frame: Up to 1 month after Multigam 5% infusion
Measure: Mean (95% Confidence Interval); unit: hour
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
hour
  Multigam 5% infusion | 4.92 [4.54 to 5.3]
  Multigam 10% infusion | 2.29 [1.96 to 2.62]
Statistical Analysis 1: Comparison: All Study Participants; H0: No difference between Multigam 5% and Multigam 10% infusion time Ha: Multigam 10% infusion time is significantly shorter than Multigam 5%; Test type: Superiority; p < 0.0001, t-test, 1 sided

2. Secondary Outcome: Hospitalisation Time of Multigam IV 5% and Multigam IV 10%
Description: Comparison of hospitalisation time (time spent at day clinic) between Multigam IV 5% and Multigam IV 10%. Results will be assessed by Student's-t-test and 95% confidence interval.
Time Frame: Up to 1 month after Multigam 5% infusion
Measure: Mean (95% Confidence Interval); unit: hour
Groups:
- All Study Participants: 30 participants who received Multigam 5% intravenous immunoglobulin (IVIg) and Multigam 10% intravenous immunoglobulin (IVIg) 3 to 4 weeks later.
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
hour
  Multigam 5% infusion | 5.87 [5.5 to 6.24]
  Multigam 10% infusion | 4.56 [3.84 to 5.27]
Statistical Analysis 1: Comparison: All Study Participants; H0: No difference in hospitalisation time between Multigam 5% and Multigam 10% infusion Ha: Hospitalisation time with Multigam 10% infusion is significantly shorter than with Multigam 5%; Test type: Superiority; p < 0.0005, t-test, 1 sided

3. Secondary Outcome: IVIg-related Adverse Events Per Patient During Multigam IV 5% and Multigam IV 10% Administration
Description: Evaluation of the occurence of adverse events (AEs) for both administrations via CTCAE v4.03 criteria.
  Results are reported as the mean number of IVIg-related AEs per patient. Adverse events were actively monitored during infusion and patients could report adverse events up to 72h after infusion.
Time Frame: Up to 72 after each infusion
Measure: Mean (95% Confidence Interval); unit: IVIg-related AEs per patient
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
IVIg-related AEs per patient
  Multigam 5% infusion | 0 [0 to 0]
  Multigam 10% infusion | 0.43 [0.12 to 0.74]

4. Secondary Outcome: Nursing Actions Per Patient During Multigam IV 5% and Multigam IV 10% Administration
Description: Evaluate the number of actions taken by the nursing staff during Multigam administration. Nursing actions were defined as the sum of actions required to increase the infusion rate (if needed) and any other action that had to be taken due to adverse effects during administration (e.g. lowering of infusion rate or supportive medication). Standard procedures like taking parameters were not accounted for this evaluation.
Time Frame: During each infusion (up to 1 day)
Measure: Mean (95% Confidence Interval); unit: Nursing actions per patient
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
Nursing actions per patient
  Multigam 5% infusion | 1.03 [0.97 to 1.1]
  Multigam 10% infusion | 0.67 [0.3 to 1.04]
Statistical Analysis 1: Comparison: All Study Participants; H0: No difference in number of nursing actions per patient between Multigam 5% and Multigam 10% infusion Ha: Number of nursing actions per patient is smaller with Multigam 10% infusion; Test type: Superiority; p = 0.03, t-test, 1 sided

5. Secondary Outcome: Patient Satisfaction Questionnaire.
Description: Assess patient satisfaction via questionnaires. Questionnaires were taken at the end of MG 10% infusion and were validated by the principal investigator (PI) and head nurse.
  Patients could score following questions from 1 (strongly disagree) to 5 (strongly agree) [Full scale: 1: strongly disagree; 2:disagree; 3: neutral; 4: agree; 5; strongly agree]:
  Question 1: I experienced less side effects during Multigam 10% infusion. Question 2: I experienced time gain with Multigam 10%. Question 3: I had a more productive day with Multigam 10%. Question 4: I am in favor of of the use of Multigam 10%.
Time Frame: End of study (after Multigam 10% infusion)
Population: Row 3: 1 patient was unable to assess the question
Measure: Median (Full Range); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
score on a scale
  Question 1 | 3 [1 to 5]
  Question 2 | 5 [2 to 5]
  Question 3: number analyzed (Participants) | 29
  Question 3 | 4 [1 to 5]
  Question 4 | 5 [1 to 5]

ADVERSE EVENTS:
Time Frame: Up to 72 after each infusion
Groups:
- Multigam 5% Infusion: 30 participants who received Multigam 5% intravenous immunoglobulin (IVIg).
- Multigam 10% Infusion: 30 participants who received Multigam 10% intravenous immunoglobulin (IVIg) 3 to 4 weeks after their Multigam 5% infusion.
Arm/Group | Multigam 5% Infusion | Multigam 10% Infusion
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 8/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multigam 5% Infusion (N=30) | Multigam 10% Infusion (N=30)
Headache (General disorders) | 0 | 4 (4)
Fatigue (General disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 1 (1) — Nausea
Infusion related reaction (General disorders) | 0 (0) | 3 (3) — Chills
Infusion related reaction (General disorders) | 0 (0) | 2 (2) — Fever

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT03250845/Prot_SAP_000.pdf